CLINICAL TRIAL: NCT06327776
Title: Nuevos Biomarcadores y Tecnologia Para Una Mejores Reglas de predicción en el Traumatismo craneoncefálico Leve
Brief Title: New Protein Biomarkers and Technology for Improving Diagnosis and Outcome Prediction in Mild TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Other Study IDs: 21/709
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-10

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MILD TBI Diagnostic and long term prognostic study: 1000 patients suffering mild Traumatic Brain Injury
  Interventions: Other: Serum and saliva biomarkers

INTERVENTIONS:
Other: Serum and saliva biomarkers — 2x5mL blood samples and saliva samples will be used to determine the performance of different blood based and saliva biomarkers for determining diagnostic management and prognosis in mTBI patients.

SUMMARY:
Mild traumatic brain injury(mTBI) is a common cause of consultation to the emergency rooms worldwide and is the most common form of traumatic brain injury. Though classified as mild, as many as 40% of patients suffering mTBI do not make complete recoveries or present persistent symptoms. The present study is intended to determine long term outcome of patients suffering mTBI and to establish new prognostic models with the use of serum and saliva based biomarkers. For this purpose this study will not exclude patients regarding their comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI (GCS 13-15 on admission)
* Blood sample obtained ≤24h after injury

Exclusion Criteria:

* GCS 3-12 on admission
* Time of injury unknown
* Time to injury exceeding 24 hours
* Primary admission for non-traumatic neurological disorder (e.g., stroke, spontaneous, intracranial hematoma)
* Penetrating head trauma
* Patient with mechanical ventilation from the trauma scene or prehospital management.
* Venipuncture not feasible
* Subject under judiciary control

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 participants suffering mild TBI
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers diagnostic performance | 24 hours after mild TBI
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of GFAP and UCHL-1, S100B, Osteopontin, SAA1, YKL-40, Copeptin, NSE, C reactive protein, procalcitonin to detect the presence or absence of intracranial lesions on CT scan

SECONDARY OUTCOMES:
Determination of the potential of the biomarkers in predicting neurological symptoms after TBI | 1 week, 3 months, 6 months and 1 year
  Early and midterm biomarker predictive performance in terms of predicting neurological outcome. Neurological status at 1 week, 3 months, 6 months and 1 year after TBI and Rivermead post concussion questionnaire.
Determination of the potential of the biomarkers in predicting neurological outcome assessed by the Extended Glasgow Outcome Score (GOSE) after TBI | 1 week, 3 months, 6 months and 1 year
  Early, midterm and long term biomarker predictive performance in terms of predicting neurological outcome. Extended Glasgow Outcome Score (GOSE)
Determination of the potential of the biomarkers in predicting quality of life assessed by Qolibri-OS after TBI | 1 week, 3 months, 6 months and 1 year
  Early, midterm and longterm biomarker predictive performance in terms of predicting quality of life after mild TBI assessed by Qolibri-OS
Determination of the potential of the biomarkers in predicting quality of life assessed by EQ-5D-5L after TBI | 3 months, 6 months and 1 year
  Mid and longterm biomarker predictive performance in terms of predicting quality of life after mild TBI assessed by EQ-5D-5L
Determination of the potential of the biomarkers in predicting quality of sleep assessed by the Epworth and Pittsburgh Scales | 3 months, 6 months and 1 year
  Mid and longterm biomarker predictive performance in terms of quality of sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No